CLINICAL TRIAL: NCT00286624
Title: A One-Year, Single-Center, Prospective, Open-Label Study of the Safety, Tolerability, and Preliminary Efficacy of Anti-Thymocyte Globulin, Cyclosporine, and RAD in Type 1 Diabetic Islet Transplant Recipients
Brief Title: Anti-Thymocyte Globulin, Cyclosporine, and RAD in Islet Transplantation
Acronym: NITA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institutes of Health (NIH) (NIH); Novartis (Industry)
Responsible Party: Bernhard J. Hering, M.D., University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0207M29841
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Everolimus; Antilymphocyte Serum; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Allogeneic islet transplantation with anti-thymocyte globulin induction and cyclosporine and RAD maintenance immunosuppression
  Interventions: Biological: Allogeneic Islets of Langerhans; Drug: Everolimus; Drug: anti-thymocyte globulin; Drug: Cyclosporine

INTERVENTIONS:
Biological: Allogeneic Islets of Langerhans — Up to 3 intraportal infusions of cadaveric pancreatic islets of Langerhans. First infusion to contain at least 5,000 islet equivalents/kg body weight. Subsequent infusions to contain at least 3,000 islet equivalents/kg body weight.
  Other Names: Islets
Drug: Everolimus — Loading dose of 3 mg PO on day -2 relative to transplant, followed at least 12 hours later by dose of 1.5 mg PO BID. The daily dose will be adjusted according to the whole blood 12-hr trough to target 3-15 ng/ml for the first 3 months and 3-12 ng/ml thereafter.
  Other Names: RAD
Drug: anti-thymocyte globulin — A total of 6 mg/kg IV over 12 hours on days -2, -1, 0, +1, and +2. The dose will be 0.5 mg/kg on day -2, 1.0 mg/kg on day -1, and 1.5 mg/kg on days 0, +1, and +2.
  Other Names: ATG; Thymogloblin
Drug: Cyclosporine — Cyclosporine started on day +1 relative to the first islet transplant. Initial dose of 3 mg/kg/day administered in 2 divided doses; then adjusted to maintain target levels of 400 (350-500) ng/mL for the first three months following islet transplant and 300 (200-350) ng/mL thereafter.
  Other Names: Neoral

SUMMARY:
This study was designed to test the safety and efficacy of up to 3 pancreatic alloislet transplants in type 1 diabetic patients with hypoglycemia unawareness. 6 subjects were transplanted under this protocol using anti-thymocyte globulin induction immunosuppression and everolimus with cyclosporine maintenance immunosuppression.

DETAILED DESCRIPTION:
This is a Phase I/II study designed to assess the safety and efficacy of sequential islet allotransplantation for the reestablishment of stable glycemic control in type 1 diabetic recipients. A total of 6 patients with type 1 diabetes have received up to three transplants of islets from different donor pancreases.

Potential candidates for islet allotransplantation included patients age 18 and older with type 1 diabetes. Induction immunotherapy for the first transplant consisted of anti-thymocyte globulin; basiliximab was used for any subsequent transplants. Peritransplant anti-inflammatory treatment with etanercept was given for each islet transplant. Maintenance immunosuppression is with cyclosporine and RAD. It is felt that those patients in whom metabolic lability/instability, reduced awareness of hypoglycemia, poor glycemic control, and progressive secondary complications persist despite continued and intensive efforts made in close cooperation with their diabetes care team are particularly likely to have a favorable benefit/risk ratio.

Adverse events, irrespective of their presumed relationship to the transplantation of allogeneic islets and/or protocol-regulated treatment products (concomitant therapy), are being monitored and recorded throughout the first year after the final islet transplant.

The proportion of single and sequential donor islet allograft recipients with full (insulin independence and HbA1c <7%) and partial (insulin dependence, basal or arginine-stimulated C-peptide levels of greater or equal to 0.5 ng/mL and HbA1c <7%) islet graft function at one year after the final islet transplant will be assessed. The impact of islet transplantation on quality of life will also be assessed.

The predictive value for posttransplant insulin independence of factors such as insulin resistance before and at intervals after pancreatectomy, cellular composition of the transplant, number of beta cells transplanted; and viability and insulin secretory response of isolated islets are being assessed.

ELIGIBILITY:
Inclusion Criteria:

* Primary islet allotransplant
* Patients with type 1 diabetes mellitus under intensive insulin management
* Age 18 or older
* Ability to give written informed consent

Exclusion Criteria:

* Age less than 18 years.
* BMI >26 kg/m2.
* Insulin requirement of > 50 IU per day.
* Positive C-peptide response to intravenous arginine stimulation.
* Untreated proliferative retinopathy.
* Creatinine clearance < 60 ml/min/1.73 m2 for females and 70 ml/min/1.73 m2 for males.
* Serum creatinine >1.3 mg/dl for females, >1.5 mg/dl for males.
* Previous pancreas or islet transplant.
* Presence of history of panel-reactive anti-HLA antibodies >10%.
* Positive pregnancy test, or presently breast-feeding, or failure to follow effective contraceptive measures.
* Active infection including hepatitis C, hepatitis B, HIV, or TB (or under treatment for suspected TB).
* Negative screen for Epstein-Barr Virus (EBV).
* Invasive aspergillus infection within year prior to study entry.
* History of malignancy.
* Active alcohol or substance abuse
* History of non-adherence to prescribed regimens.
* Psychiatric disorder making the subject not a suitable candidate for transplantation.
* Inability to provide informed consent.
* Baseline Hgb < 11.7 g/dl in females, or < 13 g/dl in males; lymphopenia (<1,000/microL), or leukopenia (<3,000 total leukocytes/microL), or an absolute CD4+ count <500/microL., or platelets <150,000/microL
* History of coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or patient with INR >1.5.
* Severe co-existing cardiac disease.
* Baseline liver function tests outside of normal range or history of significant liver disease.
* Active peptic ulcer disease.
* Severe unremitting diarrhea or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications.
* Presence of severe allergy requiring acute or chronic treatment, or hypersensitivity to drugs similar to RAD (e.g., macrolides).
* Known hypersensitivity to rabbit proteins.
* Hyperlipidemia (fasting LDL cholesterol > 130 mg/dl, treated or untreated; and/or fasting triglycerides > 200 mg/dl).
* Addison's disease.
* Under treatment requiring chronic use of systemic steroids.
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
• The incidence, timing, and severity of adverse events during one year after the first and any subsequent islet transplants. | 1 year
• Incidence and severity of hypoglycemia during the first year after the first and any subsequent islet transplants. | 1 yr
• The proportion of recipients who develop alloantibodies directed at islet donor alloantigens during the first year after the first and any subsequent islet transplants. | 1 year

SECONDARY OUTCOMES:
• The proportion of subjects who achieve insulin independence in the first year after single-donor or sequential transplantation. | 1 year
• The proportion of islet allograft recipients with full and partial islet graft function at one year after the most recent islet transplant. | 1 year
• Glycemic control and insulin secretory responses during the first year after the first and any subsequent transplants. | 1 year
• The effect of donor age, pretransplant islet insulin secretory response in vitro, number of transplanted islet equivalents (IEQ), number of transplanted beta cells, pretransplant recipient insulin requirements and action, recipient body mass index (BM | Day of transplant
• The impact of islet transplantation on the quality of life of transplant recipients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard J. Hering, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Diabetes Institute for Immunology and Transplantation - U of M — http://www.diabetesinstitute.org